CLINICAL TRIAL: NCT00075556
Title: Phase II Study Of Radiotherapy And Capecitabine As Pre-Operative Treatment In Patients With Colorectal Cancer
Brief Title: Neoadjuvant Radiation Therapy and Capecitabine in Treating Patients With Stage III or Stage IV Colorectal Adenocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000346895; FRE-GERCOR-R01-01; EU-20329
Record Dates: First submitted 2004-01-09; First posted 2004-01-12 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2008-05

CONDITIONS: Colorectal Cancer
Keywords: stage III colon cancer; stage IV colon cancer; stage III rectal cancer; stage IV rectal cancer; adenocarcinoma of the rectum; adenocarcinoma of the colon
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Capecitabine; Neoadjuvant Therapy; Radiotherapy

INTERVENTIONS:
Drug: capecitabine
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy, such as capecitabine, use different ways to stop tumor cells from dividing so they stop growing or die. Combining radiation therapy with chemotherapy before surgery may shrink the tumor so that it can be removed.

PURPOSE: This phase II trial is studying how well neoadjuvant radiation therapy and capecitabine work in treating patients who are undergoing surgery for stage III or stage IV colorectal adenocarcinoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the objective tumor response rate in patients with stage III or IV colorectal adenocarcinoma treated with neoadjuvant radiotherapy and capecitabine.

Secondary

* Determine the tolerance profile of this regimen in these patients.
* Determine the rate of preservation of functional integrity of the anal sphincter in patients treated with this regimen.
* Compare the conversion rate from the effects of mutilating surgery vs surgery with sphincter preservation in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive oral capecitabine twice daily and undergo concurrent radiotherapy 5 days a week on weeks 1-5. Patients undergo surgery on week 6.

Patients are followed every 4 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 48 patients will be accrued for this study within 10 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed colorectal adenocarcinoma

  * Clinical stage T3, T4, N+
* Measurable disease
* Awaiting surgery and likely to benefit from neoadjuvant radiotherapy

PATIENT CHARACTERISTICS:

Age

* 18 to 80

Performance status

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 2,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST and ALT no greater than 2.5 times ULN
* No hepatic condition that would interfere with study medication

Renal

* Creatinine clearance at least 80 mL/min
* No renal condition that would interfere with study medication

Cardiovascular

* No serious cardiac failure with the past year
* No myocardial infarction within the past year
* No cardiac insufficiency
* No angina
* No uncontrolled arrhythmia
* No uncontrolled hypertension

Gastrointestinal

* No superior intestinal tract malfunction
* No malabsorption syndrome

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No concurrent serious infection
* No other serious illness
* No other malignancy within the past 5 years except curatively treated basal cell skin cancer or carcinoma in situ of the cervix
* No metabolic condition that would interfere with study medication
* No dementia or altered mental status
* No psychiatric illness that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for colorectal cancer

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy for colorectal cancer

Surgery

* Not specified

Other

* More than 30 days since prior participation in another clinical study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-01

PRIMARY OUTCOMES:
Objective tumor response rate

SECONDARY OUTCOMES:
Tolerability
Rate of preservation of functional integrity of the anal sphincter
Comparison of the conversion rate from the effects of mutilating surgery vs surgery with sphincter preservation

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Dupuis, MD — Centre Jean Bernard
Locations (12):
- France (12):
  - Centre Regional Francois Baclesse, Caen
  - Hopital Drevon, Dijon
  - Hopital Saint - Louis, La Rochelle
  - Centre Jean Bernard, Le Mans
  - Clinique Saint Jean, Lyon
  - Hopital Notre-Dame de Bon Secours, Metz
  - Intercommunal Hospital, Montfermeil
  - Centre Hospitalier de Mulhouse, Mulhouse
  - Hopital Saint-Louis, Paris
  - Hopital Tenon, Paris
  - C.H. Senlis, Senlis
  - Centre Medico-Chirurgical Foch, Suresnes

REFERENCES:
- [Result] Dupuis O, Vie B, Lledo G, Hennequin C, Noirclerc M, Bennamoun M, Jacob JH. Preoperative treatment combining capecitabine with radiation therapy in rectal cancer: a GERCOR Phase II Study. Oncology. 2007;73(3-4):169-76. doi: 10.1159/000127383. Epub 2008 Apr 16. PMID 18418009